CLINICAL TRIAL: NCT01934777
Title: Study of Efficacy and Tolerance of Treatment With DHA, Choline and Vitamin E in Children With Non-alcoholic Steatohepatitis
Brief Title: Efficacy and Tolerance of Treatment With DHA, Choline and Vitamin E in Children With Non-alcoholic Steatohepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Valerio Nobili, Head of Hepato-Metabolic Disease Unit, Bambino Gesù Children Hospital, IRCCS, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPBG-DHA, VIT E, CHOLINE
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Fatty Liver; Liver Fibrosis; Obesity; Metabolic Syndrome; Nonalcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; fibrosis
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis; Obesity; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — Docosahexaenoic Acids; Vitamin E; Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TREATED GROUP (Experimental): DHA 250 mg plus Vitamin E (39 UI) plus Choline 201 mg by mouth every day in association with lifestyle intervention [hypocaloric diet (25-30 Kcal/kg/day) or isocaloric (40-45 Kcal/kg/day) and physical activity] for 6 months
  Interventions: Drug: Docosahexaenoic Acid plus Vitamin E plus choline
- PLACEBO GROUP (Placebo Comparator): placebo: this group will treated with identical placebo pearls given orally in association with lifestyle intervention [hypocaloric diet (25-30 Kcal/kg/day) or isocaloric (40-45 Kcal/kg/day) and physical activity] for 6 months
  Interventions: Drug: placebo pearls

INTERVENTIONS:
Drug: Docosahexaenoic Acid plus Vitamin E plus choline — DHA 250 mg plus Vitamin E (39 UI) plus Choline 201 mg
  Arms: TREATED GROUP
Drug: placebo pearls — placebo
  Other Names: Placebo
  Arms: PLACEBO GROUP

SUMMARY:
The purpose of this interventional study is to evaluate the efficacy and tolerability of docosahexaenoic acid (DHA), Vitamin E and Choline in children or adolescents with well-characterized and liver biopsy confirmed nonalcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
Sixty children or adolescents (4-16 years) with liver biopsy proven NAFLD will be enrolled. They will be randomized to treatment with DHA, VIT E and Choline (n=30)or an identical placebo (n=30) given orally for a period of 12 months. All patients will be included in a lifestyle intervention program consisting of a diet tailored on the individual requirements and physical exercise.

Patients will undergo a medical evaluation every three months during the 12-month study period. Liver biopsy will be performed at baseline and at 12 months. Anthropometric analysis, laboratory tests, including liver enzymes and lipids will be repeated at 3-month intervals during the 12-months study duration. Ultrasonography of the liver will be repeated after six months at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* persistently elevated serum aminotransferase levels
* diffusely echogenic liver on imaging studies suggestive of fatty liver
* biopsy consistent with the diagnosis of NAFLD

Exclusion Criteria:

* hepatic virus infections (HCV RNA-PCR negative)
* Hepatitis A, B, C, D, E and G
* cytomegalovirus and Epstein-Barr virus
* alcohol consumption
* history of parenteral nutrition
* use of drugs known to induce steatosis or to affect body weight and carbohydrate metabolism
* autoimmune liver disease, metabolic liver disease, Wilson's disease, and a-1-antitrypsin-associated liver disease were ruled out using standard clinical, laboratory and histological criteria

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Improvement in NAFLD Activity Score (NAS) | 12 months

SECONDARY OUTCOMES:
Improvement of serum alanine transferase levels, lipid profile, glico-insulinemic profile (all parameters of metabolic syndrome) and bright liver at ultrasonography | 6 and 12 months

OTHER OUTCOMES:
Safety | 6 and 12 months
  clinical examination, medical history and specific laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Valerio Nobili, MD, Principal Investigator — Bambino Gesù Children Hospital
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Rome, Italy, Italy